CLINICAL TRIAL: NCT06161389
Title: Applied Forces During Neonatal Face Mask Ventilation With Different Face-mask Air Cushion
Brief Title: Applied Forces During Neonatal Face Mask Ventilation With Different Face-mask Air Cushion Volumes
Acronym: ForVol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD3(2023)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Positive Pressure Ventilation; Preterm Infants; Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially inflated mask (Experimental): Participants will be invited to administer positive pressure ventilation by using a partially inflated mask in a neonatal manikin
  Interventions: Device: Partially inflated mask
- Fully inflated mask (Active Comparator): Participants will be invited to administer positive pressure ventilation by using a fully inflated mask in a neonatal manikin
  Interventions: Device: Fully inflated mask

INTERVENTIONS:
Device: Partially inflated mask — Manikin ventilation with a partially inflated mask
  Arms: Partially inflated mask
Device: Fully inflated mask — Manikin ventilation with a fully inflated mask
  Arms: Fully inflated mask

SUMMARY:
Positive pressure ventilation (PPV) is the most important intervention in neonatal resuscitation. During PPV, it is important to hold the face-mask with care, as applying excessive pressure could cause injury to the infant, while insufficient pressure could be a contributor of mask leak and reduced effective ventilation. Application of positive pressure to face structures may trigger a vagally mediated reflex via the trigeminal nerve that innervates the skin of the face leading to apnoea and a decrease in heart rate (TCR, trigeminal-cardiac reflex).

In neonatal manikins, ventilation with a partially or fully inflated face mask does not seem to result in differences in mask leak. The force exerted by providers to improve mask seal might result in pressure lesions and in the elicitation of the trigeminal-cardiac reflex. However, information about the applied forces is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU consultants and pediatric residents

Exclusion Criteria:

* None

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Applied forces on the manikin face | 1 minute
  The forces applied by the participants to the manikin face will be measured by sensors positioned on the manikin face

SECONDARY OUTCOMES:
Cuff pressure | 1 minute
  The pressure inside the mask will be measured during the procedure
Percentage of ventilation time with leak less than 25% around the mask | 1 minute
  The mask leak willbe measured by using a respiratory function monitoring during theprocedure

OTHER OUTCOMES:
Participants' opinion on the procedures | 5 minutes
  Participants will be asked to rate both procedures by using a Likert scale (Likert scale from 1 lowest grade to 5 highest grade)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] Schilleman K, Witlox RS, Lopriore E, Morley CJ, Walther FJ, te Pas AB. Leak and obstruction with mask ventilation during simulated neonatal resuscitation. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F398-402. doi: 10.1136/adc.2009.182162. Epub 2010 Jun 30. PMID 20591880
- [Background] van Vonderen JJ, Kleijn TA, Schilleman K, Walther FJ, Hooper SB, te Pas AB. Compressive force applied to a manikin's head during mask ventilation. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F254-8. doi: 10.1136/archdischild-2011-300336. Epub 2011 Dec 5. PMID 22147285
- [Background] Cavallin F, Sala C, Maglio S, Bua B, Villani PE, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces with direct versus indirect laryngoscopy in neonatal intubation: a randomized crossover mannequin study. Can J Anaesth. 2023 May;70(5):861-868. doi: 10.1007/s12630-023-02402-9. Epub 2023 Feb 14. PMID 36788198